CLINICAL TRIAL: NCT01948700
Title: AMICA: Assessing the Fit of Motivational Interviewing by Cultures With Adolescents
Brief Title: Assessing the Fit of Motivational Interviewing by Cultures With Adolescents
Acronym: AMICA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not an Applicable Clinical Trial (ACT).
Sponsor: University of New Mexico (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5R01AA017878-05 (NIH); 5R01AA017878-05 (NIH)
Record Dates: First submitted 2013-09-16; First posted 2013-09-24 (Estimated); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Alcoholism
Keywords: Motivational Interviewing; Problem Drinking; Adolescents; Minority Health
MeSH Terms: conditions — Alcoholism | interventions — Motivational Interviewing; Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Brief Intervention (Other): Motivational Interviewing (MI)
  Interventions: Behavioral: Motivational Interviewing
- Standard Intervention (Other): Education
  Interventions: Other: Education

INTERVENTIONS:
Behavioral: Motivational Interviewing
  Arms: Brief Intervention
Other: Education
  Arms: Standard Intervention

SUMMARY:
Hispanic adolescents experience more severe alcohol-related consequences due to their alcohol abuse and yet significantly fewer Hispanic adolescents receive alcohol treatment, particularly among justice-involved youth. Despite the level of research that has been conducted on motivational interviewing (MI) with mainstream samples, no published studies have investigated the efficacy of this brief, individual intervention with Hispanic adolescents. The overarching objective of this application is to evaluate the efficacy of a brief individual intervention (MI) for problem drinking behaviors with a sample of justice-involved Hispanic and Caucasian adolescents to determine if this intervention is differentially effective between Hispanic and Caucasian adolescents. Specifically, the first aim is to determine whether an MI intervention targeting alcohol abuse is effective at reducing alcohol use and related risk behavior in a sample of adolescent alcohol abusers. The second aim is to examine whether the effects of MI on problem drinking outcomes (e.g., alcohol problems, quantity of drinking, frequency of binging) are different between Hispanic versus Caucasian adolescents. Because it is important to determine the mechanisms that mediate the effects of MI and determine whether these mechanisms differ between Caucasian and Hispanic adolescents, the third aim is to examine whether group (Hispanic vs. Caucasian) moderates the mediational linkages in the overall model using a cross-groups approach to moderated mediation. To accomplish these aims, 453 Caucasian and Hispanic justice-involved alcohol abusing adolescents (ages 14-17) will be randomized to either two 60 minute MI interventions (one at baseline and a second, one week later) or an education condition. All adolescents will receive behavioral assessments at baseline, 3, 6 and 12 months. The proposed research is expected to take a significant step towards reducing current racial/ethnic health disparities in alcohol treatment for Hispanic adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Age 13 - 18
* Provision of informed assent (or self-consent if age 18)
* Parent/ guardian consent if under age 18
* Regular substance use (use at least 1 per month for past 6 months)

Exclusion Criteria:

* active psychosis
* mental retardation
* neurodevelopmental disorder
* severe medical illness

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 506 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Frequency of alcohol use | Change from baseline in frequency of alcohol use at 3 , 6 , & 12 month follow-up

SECONDARY OUTCOMES:
Quantity of alcohol use | Change from baseline in quantity of alcohol use at 3 , 6 , & 12 month follow-up

OTHER OUTCOMES:
Number of alcohol-related problems as indicated in the Rutgers Alcohol Problems Index | Change from baseline in number of alcohol-related problems at 3 , 6 , & 12 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Sarah W. Feldstein Ewing, Ph. D., Principal Investigator — Assistant Professor UNM
Locations (1):
- University of New Mexico Center on Alcoholism, Substance Abuse, and Addictions, Albuquerque, New Mexico, United States

REFERENCES:
- [Derived] Feldstein Ewing S, Bryan AD, Dash GF, Lovejoy TI, Borsari B, Schmiege SJ. Randomized controlled trial of motivational interviewing for alcohol and cannabis use within a predominantly Hispanic adolescent sample. Exp Clin Psychopharmacol. 2022 Jun;30(3):287-299. doi: 10.1037/pha0000445. Epub 2021 Mar 22. PMID 33749294